CLINICAL TRIAL: NCT05292599
Title: Effect of a Home-based Versus Supervised Exercise Program in Patients With Migraine: a Randomized Clinical Trial
Brief Title: Effect of a Home-based Versus Supervised Exercise Program in Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Fernando Imaz, Principal investigator, University of Gran Rosario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE versus SE in Migraine
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Migraine; Exercises
Keywords: Craniocervical flexion exercises; Neck exercises; Axioscapular exercises
MeSH Terms: conditions — Migraine Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised (Experimental): All participants in this arm will receive physiotherapy treatment that includes craniocervical flexion exercise (CCFE), isometric flexion exercises (IFE), isometric extension exercises (IEE), self-resistance exercise for neck flexion and extension (RFE), self-resistance exercise for neck rotation (RRE), midscapular exercise (ME) in 2 sessions for week, 60 minutes each, for 8 weeks. CCFE will focus on the recruitment of the deep cervical flexor muscles and will be performed from lower to higher complexity. Each of the exercises will be for 3 sets of 10 repetitions with 10 seconds of isometric contraction during the 8 weeks. IFE and IEE consist of 3 sets of 8 repetitions with 6 seconds of isometric contraction, for 6 weeks. For self-resistance exercises, the patient performs RFE and RRE. These exercises will be performed with 3 sets of 8 repetitions with 6 seconds of isometric contraction during the 8 weeks. The ME will be performed in 3 sets of 8 repetitions during the 5 weeks.
  Interventions: Other: Experimental
- No supervised (Active Comparator): The participants will perform the same exercises as the supervised group. However, in this arm will be instructed to perform the same exercises as the experimental group at home, without any supervision. These instructions will be given by the physiotherapist through videos and/or photos.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — CCFE will be performed with the patient in a supine position with both knees flexed at 45°. This exercise involves a craniocervical movement. The IFE will be performed with the patient in a supine position while the IEE will be performed in a prone position. Both exercises will activate cervical muscles. RFE and RRE will be performed with the patient in a sitting or standing position at the same time he resists with his hands on his head. ME the function of these exercises is to depress and stabilize the scapula.
  Arms: Supervised
Other: Control — CCFE will be performed with the patient in a supine position with both knees flexed at 45°. This exercise involves a craniocervical movement. The IFE will be performed with the patient in a supine position while the IEE will be performed in a prone position. Both exercises will activate cervical muscles. RFE and RRE will be performed with the patient in a sitting or standing position at the same time he resists with his hands on his head. ME the function of these exercises is to depress and stabilize the scapula.
  Arms: No supervised

SUMMARY:
Migraine is a common primary headache with documented impacts on the patient, the economy, and society. A growing number of studies have reported that people with migraines are more likely to experience neck pain and neck dysfunction. The coexistence of migraine and neck pain is also associated with a higher frequency of migraine attacks, greater susceptibility to certification. It has been reported that they present decreased cervical mobility, as well as decreased strength, resistance, and coordination of the cervical musculature of the skull. The objective of this study is to evaluate the possible clinical effects in migraineurs of supervised craniocervical and axioscapular exercises versus home-based exercises.

DETAILED DESCRIPTION:
This study will aim to verify the effect of home versus supervised exercise programs in migraine patients. The primary outcomes will be changes in the Visual Analog Scale (VAS) (0-10) and Migraine Disability Assessment Scores (MIDAS). Secondary outcomes will be changes in cervical range of motion; change in muscle endurance test; neck disability index (NDI), Headache Impact Test (HIT-6) score, Patient Health Questionnaire (PHQ-9) scores, Generalized Anxiety Disorder (GAD-7) scores.

Volunteers for the study will be included if they are between 18 and 55 years old, are of either sex, have been diagnosed with migraine according to the third edition of the International Classification of Headache, and have exhibited at least 3 days with migraine attacks in the previous month, then will be randomly assigned into two groups. A single therapist will administer the interventions twice a week for 8 weeks. The experimental group (supervised) will carry out a supervised exercises program twice a week in comparison with the control group (no supervised) and will carry out a home-based exercise program twice a week. These volunteers will be recruited at the University of Gran Rosario, (Rosario, Argentina). Primary and secondary outcomes will be measured at both groups' baseline and the end of the treatment. All the evaluations will be performed by a blinded physiotherapist

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of migraine according to the beta version of the third edition of the International Classification of Headache Disorders (ICHD), with or without pharmacological treatment.
* Age ranging between 18 to 55 years, both genders

Exclusion Criteria:

* Patients with neurological disorders (neuropathic pain or neurodegenerative disease),
* Whiplash associated disorders,
* Specific neck pain (radicular pain),
* Recent dental or physical therapy.
* If patients are taking medication to relieve pain during the study, they will be encouraged to report it.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) | At baseline and eighth weeks
  VAS is a straight horizontal line of fixed length, usually 100mm. It is a tool to assess the intensity of pain. Patients should mark their pain assessment on a scale indicated by a straight line from 0 (no pain) to 100 (pain of greatest intensity). The values will be recorded in millimeters, taken with a ruler hidden from the patient.
Change in MIDAS Scale (Migraine Disability Assessment Scale) | At baseline and eighth weeks
  The Migraine Disability Assessment (MIDAS) questionnaire is a brief, self-administered questionnaire designed to quantify headache-related disability over 3 months. Is the most widely used instrument to assess the degree of disability of patients. The disability that causes the headache is measured based on 5 questions that cover both the workplace and the domestic and family partner. Your score is obtained from the sum of the days lost by headache recorded in each of these activities, which translates into an explicit measure of time lost due to illness. This scale has shown that it is highly reliable, reproducible (regardless of the population groups evaluated), disease-specific and easy to rate, in addition to showing good internal consistency, high reliability and validity.

SECONDARY OUTCOMES:
The Cervical Disability Index (IDC) | At baseline and eighth weeks
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. It is made up of 10 elements that measure the influence of neck pain on daily activities. Individual items are scored and the total score can range from 0 to 50. Neck disability is classified as follows, based on the NDI score: 0-4 = no disability; 5-14 = mild; 15-24 = moderate; 25-34 = severe; 35 or higher = complete
The Headache Impact Test-6 (HIT-6) | At baseline and eighth weeks
  The Headache Impact Test-6 (HIT-6) was developed to measure a broad spectrum of factors that contribute to headache burden and is useful in generating quantitative and relevant information on the impact of headache. The HIT -6 is a self-reported questionnaire consisting of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five answers: "never", "rarely", "sometimes", "very often" or "always".
Neck muscle strength | At baseline and eighth weeks
  will be measured with a hand dynamometer in conjunction with a non-elastic belt to resist movement of the head, rather than the examiner's hand, to avoid any additional force from the examiner's stabilization. Neck movements included flexion, extension, and right and left lateral flexion.
Cervical flexion rotation test (FRT) | At baseline and eighth weeks
  The cervical rotation flexion test will be performed through the Easy Angle, this is an electronic goniometer, an innovative device that allows cervical mobility to be measured. This provides accurate measurements of joint mobility, is easy to use and can also save measurement results.
Patient Health Questionnaire (PHQ-9) | At baseline and eighth weeks
  This easy-to-use patient questionnaire is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the nine criteria. Where "0" (nothing) to "3" (almost every day). It has been validated for use in primary care. It is not a screening tool for depression but is used to monitor the severity of depression and response to treatment. However, it can be used to make a tentative diagnosis of depression in populations at risk.
Generalized Anxiety Disorder Assessment (GAD-7) | At baseline and eighth weeks
  This easy-to-use self-administered patient questionnaire is used as a screening tool and severity measure for generalized anxiety disorder (GAD). The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all, 'several days', 'more than half the days', and 'nearly every day, respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate, and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Numeric Pain Rating Scale | At baseline and eighth weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Imaz, PT/MSc, Principal Investigator — University of Gran Rosario
Locations (1):
- Cuadi- Universidad Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: No